CLINICAL TRIAL: NCT02228616
Title: A Multicenter, Single-Arm, Interventional, Phase 4 Study to Evaluate the Efficacy and Safety of Prucalopride in Combination With PEG or Lactulose in Women With Chronic Constipation (CC)
Brief Title: Efficacy and Safety of Prucalopride in Combination With Polyethylene Glycol or Lactulose in Women With Chronic Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR102381; PRUCOP4005 (Other: Xian-Janssen Pharmaceutical Ltd., China); PRU-C-13-CN-004-V02 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Constipation
Keywords: Constipation; Chronic constipation; Prucalopride; Women
MeSH Terms: conditions — Constipation | interventions — prucalopride; Polyethylene Glycols; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Prucalopride plus Polyethylene glycol or lactulose (Experimental)
  Interventions: Drug: Prucalopride; Drug: Polyethylene glycol (PEG); Drug: Lactulose

INTERVENTIONS:
Drug: Prucalopride — During the 12-week treatment phase of the study, the daily dose of 1 tablet of 2-mg prucalopride will be administrated orally before breakfast.
Drug: Polyethylene glycol (PEG) — Optimized dose of PEG will be administrated for 13 weeks (1 week run-in+12 weeks intervention).
Drug: Lactulose — Optimized dose of Lactulose will be administrated for 13 weeks (1 week run-in+12 weeks intervention).

SUMMARY:
The purpose of this study is to evaluate the efficacy of prucalopride 2 mg, given orally once daily for 12 weeks, in combination with PEG or lactulose, in treatment of women with Chronic Constipation (CC) in whom laxatives fail to provide adequate relief, as measured by the percentage of subjects with a weekly average increase of 1 or more spontaneous complete bowel movements (SCBMs) (responders) during the 12-week treatment phase as compared to the baseline.

DETAILED DESCRIPTION:
This is a multicenter, open-labeled, single-arm, interventional study to evaluate the efficacy and safety of prucalopride in real clinical practice.

It consists of 2 phases: a 1-week run-in phase, a 12 week, open-label treatment phase. Study population is women with CC who have been treated with laxatives but failed to obtain adequate relief within the preceding 6 months. Patients who meet the inclusive and without exclusive criteria will be enrolled in the study and signed an Informed Consent Form. They are instructed not to change their diet, lifestyle during the study.

At the first week of the study, subjects will continue PEG or lactulose treatment, and they will not be allowed to use any other laxatives and drugs for CC. Subjects will be required to maintain a written stool diary as well as the use of PEG and lactulose. Any drug affecting the colonic motility will be prohibited during the study. Following this run-in phase, subjects enter the 12-week open-label treatment phase. During the treatment phase, subjects will be treated for 12 weeks with prucalopride 2 mg, given orally once daily with or without breakfast in the morning. Subjects will be required to continue PEG or lactulose treatment with the same dosage as that in the run-in period. If necessary, due to intolerable side effects (ie, severe diarrhea,), dosage decrements of PEG or lactulose treatment may be made at any time or the subject could discontinue the PEG or lactulose treatment, based on investigator's judgement. Subjects will record study drug and laxative medication dosing information and information related to BMs in a daily diary throughout the study. PAC-SYM and PAC QOL questionnaires will be completed at Weeks 0, 4, 12. Subject safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for screening phase:
* Women aged 18 to 65 years, inclusive
* History of chronic constipation (CC): The subject reports, a weekly average of 2 or fewer spontaneous bowel movement (SBMs) and 1 or more of the following within the preceding 3 months before the screening visit, while symptom onset was more than 6 months before the screening visit: 1. very hard (little balls) and/or hard stools in more than 25% of BMs; 2. sensation of incomplete evacuation in more than 25% of BMs; 3. straining at defecation in more than 25% of BMs; 4. sensation of a no-rectal obstruction or blockade in more than 25% of BMs; 5. A need for digital manipulation to facilitate evacuation in more than 25% of BMs
* Subjects who has been using PEG or lactulose treatment for more than 1 week at screening
* Be a non-pregnant, non-lactating woman. Sexually active women must be post menopausal, surgically sterile, or practicing an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study. Women must have a negative serum beta-human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test immediately prior to study drug titration
* Inclusion Criteria for treatment phase: At Visit 2 (Week 0), the diary of Week -1 will be collected and examined for the presence of chronic constipation. The subject will be considered eligible for treatment phase if the following criteria are met: Number of SCBMs is 2 or fewer during the run-in phase (1 week)
* Subject had NO SBMs during the run-in phase is considered to be constipated

Exclusion Criteria:

* Potential subjects who meet any of the following criteria will be excluded from participating in the study
* Subjects in whom constipation is thought to be drug-induced
* Subjects suffering from secondary causes of CC
* Use of or intent to use disallowed medications that influence the bowel habit during the study (ie, anticholinergics [not including antihistamines], opioids, spasmolytics, prokinetics, and tricyclic antidepressants)
* Subjects with severe and clinically uncontrolled cardiovascular, liver, or lung disease, neurologic or psychiatric disorders (including active alcohol or drug abuse), cancer or acquired immune deficiency syndrome (AIDS), or other gastrointestinal or endocrine disorders
* Subjects with impaired renal function, i.e., serum creatinine >2 milligram/deciliter(>180 micromole/Liter)
* Subjects with clinically significant abnormalities of hematology, urinalysis, or blood chemistry
* Known allergies, hypersensitivity, or intolerance to prucalopride or its excipients
* Women who are pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with a weekly average increase of 1 or more Spontaneous Complete Bowel Movement (SCBM) during the 12-week treatment phase as compared to the baseline | 12 weeks

SECONDARY OUTCOMES:
Percentage of subjects with a weekly 3 or more Spontaneous Complete Bowel Movement (SCBM) during the 12-week treatment phase as compared to the baseline | 12 weeks
Percentage of subjects with a weekly average increase of 1 or more Spontaneous Complete Bowel Movement (SCBM) during the first 4 weeks treatment phase as compared to the baseline | 4 weeks
Percentage of subjects with a weekly average increase of 1 or more Spontaneous Bowel Movement (SBM), Bowel Movement (BM) during the 12-week treatment phase as compared to the baseline | 12 weeks
Average number of Spontaneous Complete Bowel Movement (SCBM) per week | 12 weeks
Average number of SBMs per week | 12 weeks
Average number of all BMs per week | 12 weeks
Percentage of BMs with normal consistency (Types 3-4 based on Bristol Stool Scale) per week | 12 weeks
Average weekly change of PEG or lactulose frequency and dosage as compared to baseline during the 12-week treatment phase | 12 weeks
Improvement of constipation symptoms and higher satisfaction as measured by subject's global assessments and PAC-SYM scores. Improvement is defined as that the mean score reduction from baseline is ≥0.2 | Baseline, 12 weeks
Improvement in physical, psychological, and emotional stress as measured by PAC QOL scores. Improvement is defined as that the mean score reduction from baseline is ≥0.3 | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (9):
- China (9):
  - Beijing
  - Binzhou
  - Chongqing
  - Hangzhou
  - Nanjing
  - Shanghai
  - Tianjin
  - Wuhan
  - Zhengzhou

REFERENCES:
- See also: A Multicenter, Single-Arm, Interventional, Phase 4 Study to Evaluate the Efficacy and Safety of Prucalopride in Combination With PEG or Lactulose in Women With Chronic Constipation (CC) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=5049&filename=CR102381_CSR.pdf